CLINICAL TRIAL: NCT02418481
Title: γδ T Cell Immunotherapy for Treatment of Breast Cancer
Brief Title: Safety and Efficiency of γδ T Cell Against Breast Cancer(Her-, er-, and pr-)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Gd T cell
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: γδ T Cell; breast cancer; her2-; er-; pr-
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): DC-CIK cells will be used against tumor cells.
  Interventions: Biological: DC-CIK
- Group B (Experimental): γδ T cells will be used against tumor cells.
  Interventions: Biological: γδ T Cell
- Group C (Experimental): Combination of γδ T cells/ DC-CIK be used against tumor cells.
  Interventions: Biological: Combination

INTERVENTIONS:
Biological: DC-CIK — DC-CIK cells will be used against tumor cells.
  Arms: Group A
Biological: γδ T Cell — γδ T cells will be used against breast tumor.
  Arms: Group B
Biological: Combination — γδ T/DC-CIK cells will be used against breast tumor.
  Arms: Group C

SUMMARY:
In this study, effects of γδT cells on human breast cancer (her2-, er-,pr-) in combination with tumor reducing surgery, for example cryosurgery going to be investigated.

DETAILED DESCRIPTION:
Breast tumor will be removed using tumor reducing surgery such as cryosurgery. PBMC of the patient will be separated from peripheral blood. After making them potential cancer killer γδ T Cell and DC-CIK, they will be infused to the patients as immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75
2. Karnofsky performance status >50
3. Diagnosis with breast tumors based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive cryosurgery, gd Tcells/ DC-CIK.
6. Life expectancy: Greater than 3 months
7. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other kinds of cancer
2. History of coagulation disorders or anemia
3. Patients with heart disease and diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reduced size of the tumors | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China